CLINICAL TRIAL: NCT07150013
Title: Rett REVOLUTION Trial: An Exploratory Evaluation of the Safety and Efficacy of Vorinostat in Rett Syndrome Using an "N of 1" Study Design
Brief Title: Rett REVOLUTION Trial: An Exploratory Evaluation of the Safety and Efficacy of Vorinostat in Rett Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Unravel Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RVL-001 Study 002; 20251104495 (Other: Instituto Nacional de Vigilancia de Medicamentos y Alimentos)
Record Dates: First submitted 2025-08-14; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Rett Syndrome
Keywords: n of 1; single blinded; interventional; rett syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose interventional arm (Experimental): 80mg/m2/day dose vorinostat
  Interventions: Drug: Vorinostat (SAHA)
- High dose interventional arm (Experimental): 160mg/m2/day dose vorinostat
  Interventions: Drug: Vorinostat (SAHA)
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorinostat (SAHA) — oral suspension
  Other Names: suberoylanilide hydroxamic acid
  Arms: High dose interventional arm; Low dose interventional arm
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The RETT REVOLUTION trial is a placebo-controlled, single-blinded, exploratory study with patients serving as their own control ("N of 1" trial design) where the safety and efficacy of vorinostat in the treatment of Rett syndrome will be evaluated. Each patient will be self-controlled in an adapted N-of-1 study design methodology by using a 4-week placebo baseline. Vorinostat dose escalation will occur every 8 weeks of daily dosing: placebo, 80mg/m2/day, 160mg/m2/day.

Key study objectives will include:

* To confirm the safety and tolerability of oral vorinostat 80mg/m2/day and 160mg/ m2/day dose levels when administered to typical Rett patients
* To identify the nature and magnitude of treatment response to vorinostat, as measured by changes in clinical and laboratory parameters indicative of trend towards benefit, as well as changes in mRNA expression (transcriptome response)
* Provide a data-driven justification for future study design and statistical analysis plan for subsequent clinical studies assessing safety and efficacy of vorinostat in Rett syndrome

DETAILED DESCRIPTION:
Unravel Biosciences, Inc. ("Unravel") proposes to develop an orally administered, once daily novel treatment for the orphan drug indication of Rett syndrome. Unravel has utilized its proprietary drug discovery platform to identify drugs having potential therapeutic value for neurodevelopmental disorders caused by gene mutations shown to have a cascading effect on other genes. Unravel's platform combines human gene regulatory network-based computational drug prediction with in vivo screening in a population-level diversity, CRISPR-edited, Xenopus laevis tadpole model of Rett syndrome.

Through use of Unravel's platform, the drug vorinostat ranked highly in predictive scoring, including when compared to trofinetide, which served as an active control in the screening evaluation (Novak, et.al., 2022). Vorinostat broadly improved both CNS and non-CNS (e.g., gastrointestinal, respiratory, inflammatory) abnormalities in a pre-clinical mouse model of Rett syndrome. Vorinostat was the first Rett syndrome treatment to demonstrate nonclinical efficacy across multiple organ systems when dosed after the onset of symptoms, and network analysis revealed a putative therapeutic mechanism for its cross-organ normalizing effects based on its impact on acetylation metabolism and post-translational modifications of microtubules, leading to the selection of vorinostat as a target candidate for further assessment in Rett syndrome.

The main hypotheses informing the goals and design of the study are as follows:

* Vorinostat is safe and tolerable when dosed in typical Rett patients at dose levels up to 160mg/m2/day
* At a molecular level, vorinostat mitigates the impact of the underlying MECP2 gene deficiency in Rett patients by restoring downstream mRNA synthesis, as measured by transcriptome data
* Vorinostat provides clinical benefit to Rett patients by reducing frequency and severity of clinical signs/symptoms and improving patient quality of life

The study is designed as an exploratory, proof of concept trial to investigate the study hypotheses as stated above and to achieve the primary goals of the trial. The study design adapts the well-known "n of 1" crossover study methodology (Guyatt, et.al., 1990, Kravitz, et.al., 2014), where each patient serves as their own control during comparative analyses of safety and efficacy. Up to 15 patients will be enrolled in the study to explore the hypothesis that vorinostat is a safe and potentially effective treatment for typical Rett syndrome.

Each patient enrolled in the study will be exposed to a 4-week placebo study phase to generate baseline data that will serve as a control as well as two active drug phases with vorinostat treatment, starting at 80mg/m2/day dosing for 8 weeks, followed by dose escalation to 160mg/m2/day for 8 weeks.

The study is designed to be single-blinded, where patients and their caregivers will not be aware of their treatment assignment in an attempt to minimize bias where practically possible, especially given the subjective nature of several of the endpoints being evaluated. Investigator, study staff, and sponsor will not be blinded to study treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ≥6 years of age and ≤ 21 years of age at time of screening
2. Has typical Rett Syndrome (RTT), based on diagnostic criteria for RTT described in Neul, et.al., 2010
3. Has documented, disease causing mutation in the MeCP2 gene
4. At time of screening, is in the post-regression phase with no degradation of ambulation, hand function, speech or communication skills in the 4 months prior to screening
5. Has been on a stable regimen of medication or non-pharmacological treatment for at least 4 weeks prior to the baseline visit; if currently taking trofinetide (Daybue), currently on stable dose for the previous 6 months before screening visit
6. Has had a stable pattern of seizure activity for 4 weeks before screening
7. Can swallow medication or can take it by gastrostomy tube
8. Can wear actigraphy data logging device on wrist or ankle
9. If of childbearing potential, must agree to use a highly effective method of contraception during the study and for 3 months after the last study drug administration (i.e., abstinence from sexual activity, hormonal contraceptives associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system)
10. Subjects or their legally authorized representative must be able to provide an informed consent and have sufficient language skill to complete caregiver assessments in the language in which the study assessments are provided

Exclusion Criteria:

1. Has another clinically significant medical condition other than those related to MeCP2 mutation (e.g. diabetes mellitus, cardiovascular disease, renal disease, respiratory disease, hematological abnormalities, malignancy)
2. Has major surgery planned during the study period
3. Pregnant or nursing women
4. Has a history of brain injury, stroke, other cerebrovascular disease or hypoxic-ischemic encephalopathy
5. Has clinically significant abnormal vital signs at screening or baseline
6. Has an abnormal ECG at screening, including clinically significant QT prolongation
7. Has a clinically significant abnormal laboratory value at screening
8. Liver disease or transaminase levels > 1.5 times the upper limit of the normal range as determined during screening
9. Has a history of malignancy of any organ system within the past 5 years before screening
10. Is participating in or has participated in another clinical trial within 30 days prior to the screening visit
11. Has been treated with growth hormone, IGF-1, or insulin within 12 weeks of baseline
12. Is taking anticoagulant therapy or other HDAC inhibitors
13. Has had any change to their medication or non-pharmacological treatment within 4 weeks prior to the baseline visit
14. Life expectancy of less than 12 months.
15. Has a history of alcoholism or drug/chemical abuse within 2 years before screening.
16. In the investigator's opinion, is inappropriate for this study for any reason

Ages: 6 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-related adverse events | 20 weeks
  Treatment-related adverse events coded by MedDRA will be compared qualitatively between low dose treatment, high dose treatment, and placebo groups.
Tolerability as measured by number of treatment discontinuations | 20 weeks
  The number of patients discontinuing treatment due to adverse events will be assessed between low dose treatment, high dose treatment, and placebo groups
Change in transcriptomic profile from baseline, as measured by RNA-seq (transcriptome biomarker analysis) | 20 weeks
  Transcriptome biomarker analysis is widely used to assess dynamic changes in biological systems in response to disease processes and applied stimuli, which cannot be captured with genomic sequencing of DNA mutations and variations. Unravel Biosciences has created a proprietary algorithm for analyzing transcriptome data, identifying underlying signatures of disease progression or recovery. The machine learned gene network approach predicted the use of vorinostat based on restoring a transcriptome signature of Rett syndrome toward a healthy state, which was confirmed preclinically and motivated this clinical trial. The same algorithm will be used to assess time-dependent changes in the transcriptome network signature, to evaluate its ability to capture clinical response data and to measure the extent of restoration of a disease signature back to a healthy state in a human relative to pre-clinical models.

SECONDARY OUTCOMES:
Change from baseline on the Rett-anchored Clinical Global Impression Improvement Scale (CGI-I) | 20 weeks
  7 point Likert scale with 1=very much improved and 7=very much worse
Change from baseline in Rett-anchored Clinical Global Impression Severity Scale (CGI-S) | 20 weeks
  7 point Likert Scale; 1=normal, 7=extremely ill
Change from baseline in Rett Syndrome Behavior Questionnaire (RSBQ) | 20 weeks
  The 45-item RSBQ is rated on a Likert 2-point scale and consists of eight subscales: general mood, breathing abnormalities, hand behaviors, repetitive face movements, body rocking and expressionless face, night-time behavior, fear/anxiety, and walking/standing, with ratings reflecting severity and frequency of symptoms. A total score, representing the sum of the 45 items (maximum score 90), and 8 subscale scores are obtained. A lower score represents lower symptom intensity.
Change from baseline in the Revised Motor Behavioral Assessment (R-MBA) | 20 weeks
  Each of the 24 assessment items are scored based on observed or recently reported severity/frequency and scored on a five-point Likert scale between 0 and 4, with higher numbers denoting higher levels of severity/frequency.
Change from baseline in the Caregiver Impression of Improvement (CareGI-I) | 20 weeks
  A 5-point Likert scale is used with the following response options: Much Improved (1); Improved (2); Unchanged (3); Worse (4); or Much Worse (5).
Reduction in frequency of seizures as measured by seizure diary | 20 weeks
  Caregiver-recorded seizure frequency, duration, and quality will be evaluated for evidence of improvement based on reduction in seizure burden
Changes in sleeping habits as measured by modified Child Sleep Habits Questionnaire (CSHQ) | 20 weeks
  A modified version of the 45-item caregiver questionnaire will be used. Items are rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week. Lower scores are suggestive of lower disease burden on sleep behavior
GI symptom measures relative to baseline using a subset of questions from the Gastrointestinal Symptom Rating Scale (GSRS) | 20 weeks
  A subset of 7 questions from the GSRS will be used in the study, each question rated on a 4 point ordinal scale, "0" representing no symptoms and "3" representing significant symptom burden. Lower scores reflect lower symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Neal I Muni, M.D., MSPH, Study Director — Unravel Biosciences, Inc.
Locations (1):
- Grupo de Investigación Clínica PECET (GIC-PECET), Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No